CLINICAL TRIAL: NCT04413448
Title: Performance of CT Parameters (SBAC-L1, Fractal Analysis) Compared to BMD (Gold Standard) to Detect Vertebral Fractures in rheumatoïd Arthritis
Brief Title: Performance of CT Parameters Compared to Bone Mineral Density to Detect Bone Fragility in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI083
Record Dates: First submitted 2020-05-07; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Osteoporosis; Rheumatoid Arthritis; Vertebral Fracture
MeSH Terms: conditions — Osteoporosis; Arthritis, Rheumatoid; Spinal Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: To evaluate the performance of CT parameters (SBAC-L1 and fractal analysis) compared to BMD (gold standard) to detect vertebral fractures in rheumatoid arthritis

DETAILED DESCRIPTION:
To evaluate the performance of scanographic bone attenuation coefficient of the first lumbar vertebra (SBAC-L1) and fractal analysis, markers of bone fragility on computed tomography (CT), compared to bone mineral density (BMD) to detect vertebral fractures in rheumatoid arthritis (RA).

Patient and methods: Rheumatoid arthritis patients followed from 2009 to 2019 in Nancy University hospital who met the 2010 ACR/EULAR criteria for RA and examined using thoraco-abdomino-pelvic CT (TAP-CT) and BMD (spine, hip) within a period of up to 2 years were included. Scanographic bone attenuation coefficient and fractal dimension of the first lumbar vertebra (SBAC-L1, FD-L1) were measured on CT. Vertebral fractures of the thoracolumbar spine were evaluated on CT according to an adaptation of Genant's scoring method.

Demographic characteristics (age, sex, smoking), clinical data (disease duration, DAS-28), biological data (C-reactive protein (CRP), RF, ACPA) and treatments (n proton pump inhibitor, corticosteroid, TNF-inhibitors (TNFi) and others biologics, calcium, vitamin D, antiresorptive agents) were collected from the complete medical record. Univariate and multivariate analysis were performed to determine if these variables were associated or not with bone fragility (vertebral fracture, SBAC-L1, FD-L1).

We evaluated the performance and diagnostic complementarity as well as optimal diagnostic thresholds of SBAC-L1, FD-L1 and BMD (gold standard) to detect vertebral fractures in these patients at risk of osteoporosis.

Intra and inter-readers reproducibilities of the scanographic screening methods (SBAC-L1, FD-L1) were also studied.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis patients followed from 2009 to 2019 in Nancy University hospital who met the 2010 ACR/EULAR criteria for RA
* Thoraco-abdomino-pelvic CT (TAP-CT) and BMD (spine, hip) within a period of up to 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients followed from 2009 to 2019 in Nancy University hospital who met the 2010 ACR/EULAR criteria for RA and examined using thoraco-abdomino-pelvic CT (TAP-CT) and BMD (spine, hip) within a period of up to 2 years were included.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Performance of SBAC-L1 to detect the presence of vertebral fracture on CT | 4 months
Performance of FD-L1 to detect the presence of vertebral fracture on CT | 4 months

SECONDARY OUTCOMES:
ROC curves to determine fracture thresholds to detect vertebral fractures on SBAC-L1( in Hounsfield Unit) | 1 month
Correlation between demographic , clinical, biologic and treatments and the presence of bone fragility (vertebral fracture, SBAC-L1, FD-L1) | 4 month
  Correlation between demographic (age, sexe, osteoporotic factors), clinical (disease duration, disease activity) biologic (CRP, ACPA, Rheumatoid Factor) and treatments (corticosteroids, biologic, DMARDs, anti-osteoporotic) and the presence of bone fragility (vertebral fracture, SBAC-L1, FD-L1)
ROC curves to determine fracture thresholds to detect vertebral fractures on FD-L1 | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Damien Loeuille, MD-PhD, Principal Investigator — +33662436967
Locations (1):
- University Hospital Nancy, Vandœuvre-lès-Nancy, Meurthe-et-Moselle, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.1007/s00774-013-0465-6
- See also: Related Info — http://link.springer.com/10.1007/s198-002-8335-4
- See also: Related Info — http://link.springer.com/10.1007/s00198-007-0532-8